CLINICAL TRIAL: NCT05109585
Title: Determinants of the Level of Anti-SARS-CoV-2 IgG ANTibodiEs After Vaccination (DANTE-SIRIO 7) Study
Brief Title: Determinants of the Level of Anti-SARS-CoV-2 IgG ANTibodiEs After Vaccination Study
Acronym: DANTE-SIRIO 7
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Collegium Medicum w Bydgoszczy (Other)
Responsible Party: Principal Investigator, Jacek Kubica, Professor, Collegium Medicum w Bydgoszczy
Other Study IDs: DANTE- SIRIO 7
Record Dates: First submitted 2021-11-04; First posted 2021-11-05 (Actual); Last update posted 2021-11-05 (Actual); Status verified 2021-11

CONDITIONS: SARS-CoV2 Infection; SARS-CoV2 Antibodies
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- participants willing to receive a 3-dose vaccination schedule: participants who received a 2-dose vaccination schedule, willing to receive a 3rd dose
  Interventions: Diagnostic Test: assessment of the anti-SARS-CoV-2 IgG antibody titer in 3-dose schedule
- participants unwilling to receive a 3rd dose of vaccination: participants who received a 2-dose vaccination schedule, unwilling to receive a 3rd dose
  Interventions: Diagnostic Test: assessment of the anti-SARS-CoV-2 IgG antibody titer in 2-dose schedule

INTERVENTIONS:
Diagnostic Test: assessment of the anti-SARS-CoV-2 IgG antibody titer in 3-dose schedule — evaluation of anti-SARS-CoV-2 IgG antibodies in patients after 2-dose vaccination schedule willing to receive a 3rd dose of vaccine
  Groups: participants willing to receive a 3-dose vaccination schedule
Diagnostic Test: assessment of the anti-SARS-CoV-2 IgG antibody titer in 2-dose schedule — evaluation of anti-SARS-CoV-2 IgG antibodies in patients after 2-dose vaccination schedule unwilling to receive a 3rd dose of vaccine
  Groups: participants unwilling to receive a 3rd dose of vaccination

SUMMARY:
Great expectations to control the pandemic are placed in vaccines against COVID-19. Currently, the four COVID-19 vaccines approved in the European Union. We have designed the study assessing the anti-SARS-CoV-2 IgG antibody titer after vaccination cycle the BNT162b2 vaccine in several time points relating these results to the COVID-19 history and severity of symptoms during the disease and after the first and second vaccine dose

DETAILED DESCRIPTION:
The study includes healthy, unselected volunteers from the staff of Antoni Jurasz University Hospital No.1 in Bydgoszcz and students of Collegium Medicum, Nicolaus Copernicus University. To meet the inclusion criteria patients will have to be vaccinated with two doses of the BNT162b2 vaccine. The assessment of the anti-SARS-CoV-2 IgG antibody titer at several time points in each participant. Fresh serum samples were used to measure SARS-CoV-2 IgG on the Siemens Atellica system (Siemens Healthineers, Erlangen, Germany). Results of SARS-CoV-2 IgG were given as U/ml, whereby the cut-off for positivity was defined as ≥1.0 U/ml.

ELIGIBILITY:
Inclusion Criteria:

* Provision of informed consent to study
* Age ≥ 18 years
* Receiving two doses of the BNT162b2 vaccine

Exclusion Criteria:

* patients who did not complete 2-dose vaccination schedule
* patients who received any other vaccine than BNT162b2
* patients considered by investigator to be unable to cooperate

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study includes healthy, unselected volunteers from the staff of Antoni Jurasz University Hospital No.1 in Bydgoszczand students of Collegium Medicum, Nicolaus Copernicus University.
  Approximately1000 adult participants are planned to be included in the study
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2021-04-20 (Actual); Primary Completion 2022-10-12 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
the anti-SARS-CoV-2 IgG antibody concentration 3 months after vaccination cycle with the BNT162b2 vaccine | 0-12 months
  evaluation of anti-SARS-CoV-2 IgG antibody concentration 3 months after 2-dose vaccination with BNT162b2 vaccine

SECONDARY OUTCOMES:
the anti-SARS-CoV-2 IgG antibody concentration 6, 9 and 12 months after two-dose vaccination cycle | 0-12 months
  evaluation of anti-SARS-CoV-2 IgG antibody concentration at particular time points in 2-dose vaccination schedule
the anti-SARS-CoV-2 IgG antibody concentration immediately before, 1 and 3 months after the third vaccine dose | 0-12 months
  evaluation of anti-SARS-CoV-2 IgG antibody concentration at particular time points after 3rd dose of vaccine
local and/or systemic adverse reactions after vaccination | 0-12 months
  verification of any adverse events occurrence based on survey filled by participants on each visit
confirmed COVID-19 after vaccination | 0-12 months
  verification of COVID-19 based on survey filled by participants on each visit

CONTACTS AND LOCATIONS:
Overall Officials: Jacek Kubica, Prof., Principal Investigator — Collegium Medicum w Bydgoszczy
Locations (1):
- Cardiology Department, Dr. A. Jurasz University Hospital, Bydgoszcz, Kuyavian-Pomeranian Voivodeship, Poland

IPD SHARING:
Plan to Share IPD: No